CLINICAL TRIAL: NCT03736954
Title: Pilot Study of ICU Doulas Providing Psychological Support Based on Positive Suggestions to Mitigate Psychological and Cognitive Sequelae of Critical Illness
Brief Title: ICU Doulas Providing Psychological Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lioudmila Karnatovskaia, assistant professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-008755
Record Dates: First submitted 2018-03-14; First posted 2018-11-09 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Illness, Critical; Anxiety; Depression; Post Traumatic Stress Disorder; Cognitive Impairment
MeSH Terms: conditions — Critical Illness; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICU doulas intervention (Experimental): specially trained ICU doulas will provide critically ill intubated patients with early psychological support on a daily basis
  Interventions: Behavioral: positive suggestion

INTERVENTIONS:
Behavioral: positive suggestion — humanization of critical care experience with positive reframing of hospital course on daily basis to eligible participants

SUMMARY:
Many patients who survive critical illness suffer from symptoms of anxiety, depression, or post-traumatic stress disorder (PTSD) after leaving the intensive care unit (ICU). Memories of frightening and delusional experiences in the ICU appear to be the strongest potentially modifiable risk factor. Research on the formation of fear and associated memories shows that if mitigating information about a traumatic event is introduced during the time between memory formation and its recall, the emotional experience of the memory can be modified in a positive manner. This means that in order to prevent mental health problems in critical illness survivors, psychological support needs to take place in parallel with medical treatment in the ICU. The Researchers hypothesize that early psychological support for the critically ill can decrease mental health morbidity in critical illness survivors. However, providing consistent psychological support intervention is a challenge for busy ICU clinicians. It is not feasible to hire behavioral medicine trained psychologists to become permanent ICU staff nationwide. Doulas, trained lay health care providers who provide emotional support to women in labor, have been identified as reliable yet affordable alternative. Given common elements of their services and our intervention, doulas are in an ideal position to administer early psychological support. The objective of this project is to refine and test a behavioral intervention to be administered in parallel with medical treatment in the ICU. This will be accomplished by training doulas in providing standardized psychological support intervention and refining the intervention based on stakeholder feedback

ELIGIBILITY:
Inclusion Criteria:

* adults (age >18) admitted to the ICU requiring intubation or vasopressors and expected to stay >48 hours.

Exclusion Criteria:

* history of dementia, mental retardation, suicide attempt, psychotic disorders such as schizophrenia, acute alcohol/substance intoxication or withdrawal, severe metabolic encephalopathy;
* patients on comfort care;
* patients not expected to survive the hospital stay
* non-English speaking, deaf or mute
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
feasibility of integration of trained doulas into the ICU | 6 months
  pilot feasibility study. Feasibility defined as ICU doulas being able to perform study intervention on 30 recruited patients for at least 10 minutes daily throughout patient's ICU course.

SECONDARY OUTCOMES:
Patient scores on Hospital Anxiety and Depression Scale | 6 months
  quantitative. Study patients will complete follow-up questionnaires measuring symptoms of anxiety and depression following ICU discharge but prior to hospital discharge. Patient's scores on these questionnaires will be compared to propensity-matched historic cohort.
Patient scores on Impact of Events Scale - Revised | 6 months
  quantitative. Study patients will complete follow-up questionnaires measuring symptoms of acute stress following ICU discharge but prior to hospital discharge. Patient's scores on these questionnaires will be compared to propensity-matched historic cohort.
Patient scores on Montreal Cognitive Assessment-blind | 6 months
  quantitative. Study patients will complete follow-up questionnaires measuring cognitive function following ICU discharge but prior to hospital discharge. Patient's scores on these questionnaires will be compared to propensity-matched historic cohort.
Qualitative interviews of patients, their family members, physicians and nurses caring for the study patients | 6 months
  We will use an "interpretive description approach" to qualitative research, which creates an interpretive account of a clinical phenomenon for the purpose of informing clinical practice. We aim to understand the changes in experiences of critically ill patients, their family members, and providers through the interviews. This allows us to explore patient and key stakeholders' perspectives and to refine PSBPS based on the areas of highest priority, focusing on elements that are deemed by patients to be of highest acceptability. Following patient ICU discharge, interviews will be conducted on a one-on-one basis by the candidate or a trained qualitative interviewer who is not directly involved in the patient's clinical care; participants will be assured that interview transcripts will be confidential. Interviews will last approximately 15 minutes and will be conducted in person.

CONTACTS AND LOCATIONS:
Overall Officials: Lioudmila V Karnatovskaia, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Karnatovskaia LV, Varga K, Niven AS, Schulte PJ, Mujic M, Gajic O, Bauer BA, Clark MM, Benzo RP, Philbrick KL. A pilot study of trained ICU doulas providing early psychological support to critically ill patients. Crit Care. 2021 Dec 20;25(1):446. doi: 10.1186/s13054-021-03856-3. PMID 34930440
- [Background] Karnatovskaia LV, Schultz JM, Niven AS, Steele AJ, Baker BA, Philbrick KL, Del Valle KT, Johnson KR, Gajic O, Varga K. System of Psychological Support Based on Positive Suggestions to the Critically Ill Using ICU Doulas. Crit Care Explor. 2021 Apr 26;3(4):e0403. doi: 10.1097/CCE.0000000000000403. eCollection 2021 Apr. PMID 33912833
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials